CLINICAL TRIAL: NCT04456790
Title: Plenvu 1 - Questionnaire Study Exploring Patients Preference in Bowel Preparation Timings for Morning Colonoscopy
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/32
Record Dates: First submitted 2020-02-19; First posted 2020-07-07 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Bowel Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Questionnaire study exploring patients preference in bowel preparation timings for morning colonoscopy.

DETAILED DESCRIPTION:
It is often difficult to achieve optimal bowel cleansing for patients having morning colonoscopies. One possible cause of this is the timing of the bowel preparation prior to the procedure. A clean bowel will allow for a clear view of its inner lining which is important for both accurate diagnosis and treatment. Abnormal changes may be tiny, so even the smallest amount of faeces could potentially disguise polyps and cancers.

Additionally, poor bowel cleansing can lead to the procedure being cancelled and repeated on another occasion at a later date, adding to the burden on current resources. Poor bowel preparation has also been shown to be a factor in more difficult and longer procedures, increased patient discomfort, and a higher risk of complications.

This is more of an issue for patients having a colonoscopy in the morning. One cause of this could be the timing of bowel preparation. Studies have shown that having a smaller window of time between finishing bowel preparation and having a colonoscopy results in a much cleaner bowel. The investigators are therefore considering the times patients are required to take their bowel preparation in order to improve the bowel cleansing outcome for a morning colonoscopy.

Previous studies have indicated that a split dose (one evening dose and one early morning dose) improves bowel cleansing compared to all doses taken the day prior to colonoscopy. However, there has been no research to assess the efficacy of early morning bowel preparation and its acceptability to patients. This information may lead to future studies and in order to ensure the success of this further research it is important to understand any potential barriers from patients to new timing regimens.

Therefore, such information as highest education level, employment status, age and experience of previous bowel preparation for colonoscopy for the patient population is captured.

Results from previous studies looking at potential barriers have shown that such issues as having a simplified colonoscopy instruction sheet improved bowel preparation and lowered cancellation rates and that patients with a history of colonoscopy are less likely to follow bowel preparation instructions and therefore achieve adequate bowel cleansing.

A total of 300 participants will be approached; 150 participants who have previously had bowel preparation for colonoscopy and 150 participants who have not, and are attending for a flexi sigmoidoscopy and therefore may have to go on to have a colonoscopy.

These groups will be further split to half attending in the morning and half attending in the afternoon, thus achieving a cross section of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* • Attending the endoscopy suite at Portsmouth Hospitals NHS Trust for colonoscopy or flexi-sigmoidoscopy procedures

  * Aged 18 years and above
  * Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* • Aged under 18 years

  * Unable to complete the questionnaire unsupervised

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients attending the endoscopy unit for a flexible sigmoidoscopy or colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Patient preferences questionnaire | 3 months
  Patients to rate their preference for timings from 1st to third choice.

SECONDARY OUTCOMES:
Patient preferences questionnaire | 3 months
  To establish the reasons for expressed preferences for bowel preparation timings

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Sr Dash, Principal Investigator — Portsmouth NHS Hosptials Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Wessex, United Kingdom

IPD SHARING:
Plan to Share IPD: No